CLINICAL TRIAL: NCT06624696
Title: Inhaling Penehyclidine to Prevent Perioperative Respiratory Adverse Events in Children at Risk Undergoing Sevoflurane Anesthesia: a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Inhaling Penehyclidine to Prevent Perioperative Respiratory Adverse Events in Children at Risk Undergoing Sevoflurane Anesthesia
Acronym: PEPSI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shenzhen Eye Hospital (Other)
Responsible Party: Principal Investigator, Xiaoliang Gan, The head of Anesthesiology, Zhongshan Ophthalmic Center, Sun Yat-sen University, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IIT2024111
Record Dates: First submitted 2024-09-30; First posted 2024-10-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Hypersensitivity; Perioperative Respiratory Adverse Events; Anticholinergics; Inhalation Therapy; Complications; High Risk
Keywords: perioperative respiratory adverse events; pediatric anesthesia; penehyclidine; sevoflurane
MeSH Terms: conditions — Respiratory Hypersensitivity | interventions — penehyclidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The penehyclidine hydrochloride group (Experimental): Inhaling penehyclidine hydrochloride (a dose of 0.05 mg/kg, diluted and mixed with normal saline to a total volume of 5 ml) for nebulization therapy within 30 min prior to surgery.
  Interventions: Drug: Penehyclidine hydrochloride
- The normal saline group (Placebo Comparator): Inhaling normal saline in a total volume of 5 ml for nebulization therapy within 30 min prior to surgery.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Penehyclidine hydrochloride — The penehyclidine hydrochloride will be diluted to a total volume of 5 mL with normal saline, added to the nebulizer cup for inhalation. Patients will be asked to inhale the entire volume of nebulized drugs within 30 min prior to surgery. The trial drugs will be administered using a jet nebulizer with compressed air flow. Each child will be intructed to begin the nebulization by using a face mask that covers the nose and mouth while the child is seated upright. Children will be encouraged to take deep and slow breaths, inhaling through the mouth and exhaling through the nose, to ensure the drugs effectively reaches the airway.
  Arms: The penehyclidine hydrochloride group
Drug: Normal Saline — The normal saline with a total volume of 5 mL will be added to the nebulizer cup for inhalation. Patients will be asked to inhale the entire volume of nebulized drugs within 30 min prior to surgery. The trial drugs will be administered using a jet nebulizer with compressed air flow. Each child will be intructed to begin the nebulization by using a face mask that covers the nose and mouth while the child is seated upright. Children will be encouraged to take deep and slow breaths, inhaling through the mouth and exhaling through the nose, to ensure the drugs effectively reaches the airway.
  Arms: The normal saline group

SUMMARY:
This randomized controlled study is to evaluate the effectiveness of inhaling penehyclidine hydrochloride in reducing perioperative respiratory adverse events in children at risk undergoing minor elective surgery.

DETAILED DESCRIPTION:
Children with high risk factors of perioperative respiratory adverse events (PRAEs) remains a challenge for general anesthesia, inhalation of penehyclidine hydrochloride (PHC) has been showed to reduce postoperative pulmonary complications and enhance the recovery in high-risk surgical patients. Thus, prophylactic PHC inhalation might show promising benefits against PRAEs in pediatric anesthesia. This clinical study is designed to test the hypothesis that pediatric patients who exist at least 1 risk factor of PRAEs prophylactically to inhale PHC have a lower prevalence of PRAEs.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients aged 3 to 7 years.
2. Scheduled to undergo ophthalmic surgery.
3. Judged to be at risk of PRAEs (with at least one parentally reported risk factor for the PRAEs, including history of a recent cold, wheezing during exercise, wheezing more than three times in the past 12 months, nocturnal dry cough, eczema, or a family history of asthma, rhinitis, eczema, or exposure to passive smoke).

Exclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical classification ≥ IV.
2. Known cardiopulmonary diseases (eg. uncorrected congenital heart disease, primary or secondary pulmonary hypertension, tumors, or structural lung diseases).
3. Severe renal dysfunction (requirement of renal replacement therapy) or severe hepatic dysfunction (Child-Pugh grade C);
4. Neurological disorders.
5. Neuromuscular diseases.
6. Contraindication for PHC.
7. Inhalation of β2-receptor activator, M-receptor blockers and/or glucocorticoids within 1 month before surgery.
8. Allergy to anticholinergic drugs.
9. Use of endotracheal tube (ETT) for ventilation.
10. Known difficult airway.
11. Severe upper respiratory tract infections (URTIs) and the anesthesiologist recommended delaying surgery.
12. Participation in other clinical trial during the last month or within the six half-life periods of the study drug used in the last trial.
13. Parents refusing to allow their children to participate.
14. Obesity, with a body mass index (BMI) over 95th percentile according to the WHO guideline.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 204 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of PRAEs | From beginning of anesthesia induction until the completion of postoperative recovery in PACU (including the phases of anesthesia induction, anesthesia maintenance, postoperative emergency and postoperative recovery), assessed up to 24 hours.
  PRAEs are subdivided into two types: major (bronchospasm and laryngospasm) and minor (severe coughing, breath holding, desaturation, upper airway obstruction, and stridor) events. The primary outcome is the incidence of PRAEs. Patients will be considered positive for respiratory adverse events if at least 1 of the above adverse events occurs.

SECONDARY OUTCOMES:
The severity of major respiratory adverse events if occurs | From beginning of anesthesia induction until the completion of postoperative recovery in PACU (including the phases of anesthesia induction, anesthesia maintenance, postoperative emergency and postoperative recovery), assessed up to 24 hours.
  Major respiratory adverse events include laryngospasm and bronchospasm. Laryngospasm will be scored according to its severity as follows: 1=none, 2=partial-reposition airway, 3=partial-continuous positive airway pressure (CPAP), 4=complete-muscle relaxant. Bronchospasm will be scored according to its severity as follows: 1=none, 2= expiration only, 3= expiration and inspiration, 4=difficult to ventilate, require treatment.
Ease of LMA insertion | From the beginning of LMA insertion until the completion of successful LMA insertion, assessed up to 24 hours
  This outcome includes time to successful insertion, the number of insertion attempts, and difficulty at insertion.
The episode and degree of salivation during removal of LMA | At the time of LMA removal, assessed up to 24 hours
  Degree of salivation is evaluated as follows: 1=none; 2=minimal, no suction; 3=moderate, suction 1×; 4=copious, suction>1×.
The airway hyperreactivity score | From the time of LMA removal until regaining consciousness from anesthesia, assessed up to 24 hours
  This score is used to assessed severity of PRAEs, accounting for the intensity of coughing, breath holding, and oxygen desaturation on a scale ranging from 0 (none) to 4 (severe). The maximum score is 12, and a score of ≤3 is categorized as mild, 4 to 8 as moderate, and ≥9 as severe.
The anesthesia-related time | During the phases of anesthesia emergence and recovery, assessed up to 24 hours
  The anesthesia-related time includes time to LMA removal, and PACU stay time.
Emergence agitation | From the time of LMA removal until regaining consciousness from anesthesia, assessed up to 24 hours
  Emergence agitation will be evaluated within stay in PACU using the Aono's four point scale (1: calm; 2: not calm but easily consolable; 3: not easily calmed restless or moderately agitated; 4: combative, disoriented, or excited). The scale scoring of 1 and 2 are considered as the absence of EA, and scale of 3 and 4 are considered as the presence of EA.
Postoperative pain score | From the time of arrival in PACU until the time of discharge from PACU, assessed up to 24 hours
  Postoperative pain score will be assessed within stay in the PACU using the Wong-Baker Pain Scale. A score higher than 4 is defined as moderate-to-severe pain which need to be timely managed.
The change of systolic blood pressure (SBP) | At baseline; 5 minutes after inhaling PHC; the completion of inhaling PHC; LMA insertion; upon arrival in PACU; pre-LMA mask removal; post-LMA mask removal; ready to discharge from PACU, assessed up to 24 hours
  The changes of SBP will be recorded.
The change of heart rate (HR) | At baseline; 5 minutes after inhaling PHC; the completion of inhaling PHC; LMA insertion; upon arrival in PACU; pre-LMA mask removal; post-LMA mask removal; ready to discharge from PACU, assessed up to 24 hours
  The changes of HR will be recorded.
The change of SpO2 | At baseline; 5 minutes after inhaling PHC; the completion of inhaling PHC; LMA insertion; upon arrival in PACU; pre-LMA mask removal; post-LMA mask removal; ready to discharge from PACU, assessed up to 24 hours
  The change of SpO2 will be recorded.
Other adverse events | From beginning of inhalation until the 24 postoperative hours.
  Other adverse events potentially related to inhale the study drug from beginning of inhalation until the 24 postoperative hours, including postoperative nausea and vomitting (PONV), dry month, palpation, dizziness, fever, cough, urine retention, and flushing.
The incidence of respiratory infections within 7 days after surgery | Within 7 days after surgery.
  Children who develop respiratory infections within 7 days after surgery will be recorded during postoperative follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen Eye Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tait AR, Malviya S, Voepel-Lewis T, Munro HM, Seiwert M, Pandit UA. Risk factors for perioperative adverse respiratory events in children with upper respiratory tract infections. Anesthesiology. 2001 Aug;95(2):299-306. doi: 10.1097/00000542-200108000-00008. PMID 11506098
- [Background] Ramgolam A, Hall GL, Sommerfield D, Slevin L, Drake-Brockman TFE, Zhang G, von Ungern-Sternberg BS. Premedication with salbutamol prior to surgery does not decrease the risk of perioperative respiratory adverse events in school-aged children. Br J Anaesth. 2017 Jul 1;119(1):150-157. doi: 10.1093/bja/aex139. PMID 28974069
- [Background] Tait AR, Voepel-Lewis T, Burke C, Kostrzewa A, Lewis I. Incidence and risk factors for perioperative adverse respiratory events in children who are obese. Anesthesiology. 2008 Mar;108(3):375-80. doi: 10.1097/ALN.0b013e318164ca9b. PMID 18292674
- [Background] An MZ, Xu CY, Hou YR, Li ZP, Gao TS, Zhou QH. Effect of intravenous vs. inhaled penehyclidine on respiratory mechanics in patients during one-lung ventilation for thoracoscopic surgery: a prospective, double-blind, randomised controlled trial. BMC Pulm Med. 2023 Sep 19;23(1):353. doi: 10.1186/s12890-023-02653-8. PMID 37726724
- [Background] Yan T, Liang XQ, Wang GJ, Wang T, Li WO, Liu Y, Wu LY, Yu KY, Zhu SN, Wang DX, Sessler DI. Prophylactic Penehyclidine Inhalation for Prevention of Postoperative Pulmonary Complications in High-risk Patients: A Double-blind Randomized Trial. Anesthesiology. 2022 Apr 1;136(4):551-566. doi: 10.1097/ALN.0000000000004159. PMID 35226725
- [Background] Wang NA, Su Y, Che XM, Zheng H, Shi ZG. Penehyclidine ameliorates acute lung injury by inhibiting Toll-like receptor 2/4 expression and nuclear factor-kappaB activation. Exp Ther Med. 2016 May;11(5):1827-1832. doi: 10.3892/etm.2016.3154. Epub 2016 Mar 11. PMID 27168812
- [Background] Wang Y, Gao Y, Ma J. Pleiotropic effects and pharmacological properties of penehyclidine hydrochloride. Drug Des Devel Ther. 2018 Oct 5;12:3289-3299. doi: 10.2147/DDDT.S177435. eCollection 2018. PMID 30323561
- [Background] Tait AR, Burke C, Voepel-Lewis T, Chiravuri D, Wagner D, Malviya S. Glycopyrrolate does not reduce the incidence of perioperative adverse events in children with upper respiratory tract infections. Anesth Analg. 2007 Feb;104(2):265-70. doi: 10.1213/01.ane.0000243333.96141.40. PMID 17242078
- [Background] Wudineh DM, Berhe YW, Chekol WB, Adane H, Workie MM. Perioperative Respiratory Adverse Events Among Pediatric Surgical Patients in University Hospitals in Northwest Ethiopia; A Prospective Observational Study. Front Pediatr. 2022 Feb 11;10:827663. doi: 10.3389/fped.2022.827663. eCollection 2022. PMID 35223702
- [Background] Ramgolam A, Hall GL, Zhang G, Hegarty M, von Ungern-Sternberg BS. Deep or awake removal of laryngeal mask airway in children at risk of respiratory adverse events undergoing tonsillectomy-a randomised controlled trial. Br J Anaesth. 2018 Mar;120(3):571-580. doi: 10.1016/j.bja.2017.11.094. Epub 2018 Jan 27. PMID 29452814
- [Background] von Ungern-Sternberg BS, Sommerfield D, Slevin L, Drake-Brockman TFE, Zhang G, Hall GL. Effect of Albuterol Premedication vs Placebo on the Occurrence of Respiratory Adverse Events in Children Undergoing Tonsillectomies: The REACT Randomized Clinical Trial. JAMA Pediatr. 2019 Jun 1;173(6):527-533. doi: 10.1001/jamapediatrics.2019.0788. PMID 31009034
- [Background] Peterson MB, Gurnaney HG, Disma N, Matava C, Jagannathan N, Stein ML, Liu H, Kovatsis PG, von Ungern-Sternberg BS, Fiadjoe JE; PAWS-COVID-19 Group. Complications associated with paediatric airway management during the COVID-19 pandemic: an international, multicentre, observational study. Anaesthesia. 2022 Mar 23;77(6):649-58. doi: 10.1111/anae.15716. Online ahead of print. PMID 35319088
- [Background] Oofuvong M, Geater AF, Chongsuvivatwong V, Chanchayanon T, Sriyanaluk B, Saefung B, Nuanjun K. Excess costs and length of hospital stay attributable to perioperative respiratory events in children. Anesth Analg. 2015 Feb;120(2):411-9. doi: 10.1213/ANE.0000000000000557. PMID 25517194
- [Background] Hii J, Templeton TW, Sommerfield D, Sommerfield A, Matava CT, von Ungern-Sternberg BS. Risk assessment and optimization strategies to reduce perioperative respiratory adverse events in pediatric anesthesia-Part 1 patient and surgical factors. Paediatr Anaesth. 2022 Feb;32(2):209-216. doi: 10.1111/pan.14377. Epub 2021 Dec 20. PMID 34897906
- [Background] Shen F, Zhang Q, Xu Y, Wang X, Xia J, Chen C, Liu H, Zhang Y. Effect of Intranasal Dexmedetomidine or Midazolam for Premedication on the Occurrence of Respiratory Adverse Events in Children Undergoing Tonsillectomy and Adenoidectomy: A Randomized Clinical Trial. JAMA Netw Open. 2022 Aug 1;5(8):e2225473. doi: 10.1001/jamanetworkopen.2022.25473. PMID 35943745
- [Background] Lin Y, Chen Y, Huang J, Chen H, Shen W, Guo W, Chen Q, Ling H, Gan X. Efficacy of premedication with intranasal dexmedetomidine on inhalational induction and postoperative emergence agitation in pediatric undergoing cataract surgery with sevoflurane. J Clin Anesth. 2016 Sep;33:289-95. doi: 10.1016/j.jclinane.2016.04.027. Epub 2016 May 18. PMID 27555179